CLINICAL TRIAL: NCT00963677
Title: Shikani Optical Stylet for Nasotracheal Intubation Undergoing Oral and Maxillofacial Surgery, a Prospective Evaluation
Brief Title: Nasotracheal Intubation Using Shikani Optical Stylet
Acronym: SOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Ru-Ping Dai, Associate Professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSFC-30700790; RDai-CSU (Other: Central South University)
Record Dates: First submitted 2009-08-19; First posted 2009-08-21 (Estimated); Results first posted 2012-05-03 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-03

CONDITIONS: Intubation; Difficult
Keywords: Shikani optical stylet(SOS); difficult airways; intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intubation without difficulty (Experimental): The patients are not predicted for difficult intubation
  Interventions: Procedure: Nasotracheal Intubation through seeing optical stylet (SOS)
- Difficult intubation (Experimental): The patients will be anticipated for difficult intubation without difficult ventilation
  Interventions: Procedure: Nasotracheal Intubation through seeing optical stylet (SOS)

INTERVENTIONS:
Procedure: Nasotracheal Intubation through seeing optical stylet (SOS) — Nasotracheal intubation using seeing optical stylet in the patients with the anticipated difficult intubation. Arm 1:routine anesthesia induction,0.1mg/kg midazolam, 3-8mcg/kg fentanyl, 0.08-0.15mg/kg vecuronium and 0.3mg/kg etomidate, Nasotracheal intubation with seeing optical shikani; Arms 2: Sevoflurane combined with oxyge, 0.3mg/kg Etomidate and 1-2mg/kg succinylcholine for intubation, nasotracheal intubation with seeing optical shikani
  Other Names: fluoroscopy

SUMMARY:
Difficult airways is still a challenging issue for the anesthesiologists in spite of the development of various techniques.Shikani optical stylet(SOS), combining the features of fiberoptic bronchoscope and a lightwand, has been used for orotracheal intubation with difficult airways. As compared with fiberoptic bronchoscope, SOS is less expensive, easy to learn and more durable. However, it remains elusive whether SOS can be used in the nasotracheal intubation in the oral and maxillofacial surgery, which normally requires the nasotracheal intubation. The present study evaluates the safety and efficacy of SOS for nasotracheal intubation in the oral and maxillofacial surgery requiring nasotracheal intubation.

DETAILED DESCRIPTION:
The present study has been approved by the Research Ethics Committee of the Second Xiangya Hospital of Central South University . Informed and written consent will be obtained from patients who are undergoing oral and maxillofacial surgery requiring general anesthesia with nasotracheal intubation. Preoperative clinical assessment of the patients will include routine airway evaluation of dentition, mouth opening, tongue size, Mallampati score, and neck mobility.

For the patients without anticipated difficult intubations. Patients will be induced by the routine anesthesia fashion including 0.1mg/kg midazolam, 3-8mcg/kg fentanyl, 0.08-.015mg/kg vecuronium and 0.3mg/kg etomidate with standard preoxygen. The patients will be ventilated with 100% oxygen via bag and mask for 3 minutes.

For the patients with anticipated difficult airways. Patients will be inhaled with sevoflurane in 100% oxygen. Some protocols will be performed as the following: 1)If the patient can be ventilated with bag and mask after losing consciousness, 0.3mg/kg etomidate and 1-2mg/kg succinylcholine will be administered for muscle paralysis. If not, sevoflurane will be stopped and the patient will be awakened. Fiberoptic bronchoscope will be performed for the intubation; 2)If two attempts of intubation with SOS are failed, then the direct laryngoscope will be used for the intubation; If the intubation with direct laryngoscope is also failed, the patients will be awakened and intubated in the awake status.

After confirmation of the successful intubation, the routine anesthesia fashion will be followed and the surgery will be performed as the usual fashion.

Intubation time will be defined as the time from when Shikani stylet passes the nose of the patient until the time the endotracheal tube is positioned in the trachea. If the intubation sequence is longer than 120 seconds, it will be deemed a failure and recorded as such.

ELIGIBILITY:
Inclusion Criteria:

* Elective non-cardiac surgery patients requiring intubation for the surgery. Age 18-70 ASA 1-3 Body Mass Index (BMI) < 40

Exclusion Criteria:

* Patients confirmed with difficult ventilation;
* Patients not suitable for nasal intubation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Ping Dai, MD, PhD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (ASA I-III) who required general anesthesia undergoing oral and maxillofacial surgery and agreed to participate in the present study were recruited from August 2009 to November 2009 in the Second Xiangya Hospital of Central South university. All the patients have signed the consented forms for the study.
Pre-assignment Details: 55 patients were recruited into the study and assigned to two groups. The patients without predicted difficult intubation (n=35) were rectuited into Group A. The patients (n=20) with predicted intubation but not difficult ventilation were recruited into Group B. Two patients were excluded from the present study due to difficult ventilation.
Groups:
- Intubation Without Difficulty: Patients without anticipated difficult intubation. Anesthesia induction: Midalozlam, Fentanyl, Vecuronium; Etomidate. After that, nasotracheal intubation with Shikani optical stylet
- Difficult Intubation: The patients will be anticipated for difficult intubation without difficult ventilation. Anesthesia was induced by inhaled sevoflurane with oxygen followed by 0.3mg/kg etomidate and 1-2mg/kg succinylcholine. After induction, nasotracheal inbutation were performed with seeing optical shikani.
Period: Overall Study
Arm/Group | Intubation Without Difficulty | Difficult Intubation
Started | 35 (Patients without predicted difficult intubation) | 20 (Patients with predicted difficult intubation but not ventilation)
Completed | 35 | 18 (Two patients were excluded from the study due to the difficult ventilation with facemask ventilation)
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intubation Without Difficulty | Difficult Intubation | Total
Number analyzed (Participants) | 35 | 20 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 20 | 55
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.2 (6.7) | 32.7 (6.3) | 33.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 20 | 11 | 31
Region of Enrollment [Number; unit: participants]
  China | 35 | 20 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of the Patients With Successful Nasotracheal Intubation
Description: After anesthesia induction, the patients were undergone nasotracheal intubation with SOS. Number for first time successful intubation was recorded. If the time for one attempt intubation exceeded more than 120 seconds, it would be regarded as failed intubation for this time intubation. If a patient could not be successfully intubated after three attempts, the patients would be viewed as a case failing nasotracheal intubation with SOS.
Time Frame: 1 hour(peri-intubation time)
Measure: Number; unit: participants
Arm/Group | Intubation Without Difficulty | Difficult Intubation
Number analyzed (Participants) | 35 | 20
participants | 35 | 18

2. Secondary Outcome: Time for Nasotracheal Intubation With the Use of Shikani Optical Stylet
Description: The time of nasotracheal intubation was calculated from the SOS insertion to withdrawing the stylet from the endotracheal tube.
Time Frame: 1 hour (peri-intubation time)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intubation Without Difficulty | Difficult Intubation
Number analyzed (Participants) | 35 | 20
seconds | 26.3 (6.4) | 27.2 (8.1)

ADVERSE EVENTS:
Arm/Group | Intubation Without Difficulty | Difficult Intubation
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/18
Other Adverse Events (participants affected / at risk) | 0/35 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes